CLINICAL TRIAL: NCT00284505
Title: Prospective Study of the Use of Thalidomide in Patients With Arachnoiditis
Brief Title: Use of Thalidomide in Patients With Arachnoiditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG0678
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Arachnoiditis
Keywords: cytokine; arachnoiditis; neuropathic pain; tumor necrosis factor
MeSH Terms: conditions — Arachnoiditis; Neuralgia | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
This pilot study will evaluate whether thalidomide decreases pain in patients with arachnoiditis.

DETAILED DESCRIPTION:
Arachnoiditis, a neuropathic disease caused by inflamation of the arachnoid membrane that surrounds and protects the spinal nerves,can result in a debilitating state that is characterized by numbing and tingling, stinging and burning in the lower back or legs, and possible muscle cramps, twitching and spasms. Current treatments are not always effective in treating the pain associated with arachnoiditis. Recent research has indicated that a group of chemicals called cytokines that are produced by various cells in the body may be responsible for generating the pain response. Medications that effect the release of cytokines or block the action of cytokines may reduce the pain response. Various anti-cytokine medications are now being used to treat painful disease states such as rheumotoid arthritis and Crohn's Disease. In this study the anti-cytokine medication, Thalidomide, is being evaluated for it's effect in treating pain associated with arachnoiditis.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically confirmed Arachnoiditis
* Involvement of the lower limb(s)

Exclusion Criteria:

* Subjects with baseline peripheral neuropathy to include diabetic neuropathy and other metabolic or toxic neuropathies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2005-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
1. To evaluate the change in pain as measured by the McGill Pain Questionnaire, short form, (SF-MPQ) and consumption of adjuvant opioid medications in three patients with arachnoiditis who receive thalidomide.
2. To evaluate the change in physical functionality as measured by the Roland-Morris Low Back Pain and Disability Questionnaire in three patients with arachnoiditis who receive thalidomide.

SECONDARY OUTCOMES:
1. To measure change in the patient's health status as measured by the SF36 in three patients with arachnoiditis who receive thalidomide.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony H Guarino, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Pain Management Center, St Louis, Missouri, United States